CLINICAL TRIAL: NCT01672905
Title: Evaluation of PSA Antibody on E9802: Confirmation and Concordance
Brief Title: PSA Antibody Levels in Samples From Patients With Prostate Cancer Treated on Protocol ECOG-E9802
Status: Completed | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000738979; ECOG-E9802T1
Record Dates: First submitted 2012-08-23; First posted 2012-08-27 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage I prostate cancer; stage IIA prostate cancer; stage IIB prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood or tumor tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

PURPOSE: This clinical trial studies prostate-specific antigen (PSA) antibody levels in samples from patients treated for prostate cancer on trial ECOG-E9802.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate changes in prostate-specific antigen (PSA) antibody levels over time among patients treated on ECOG-E9802.

Secondary

* To characterize the concordance of PSA antibody assessment between the ECOG Immunology Laboratory and the NCI Immunology Laboratory.

OUTLINE: Previously tested samples are evaluated for changes in PSA antibody levels over time (from baseline to follow-up at 12 and 24 weeks) at the ECOG Immunology Laboratory and the NCI Immunology Laboratory. Results are compared between the laboratories.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Samples collected on ECOG-E9802 (A Phase II Study of PROSTVAC-V (Vaccinia)/TRICOM and PROSTVAC-F (Fowlpox/TRICOM with GM-CSF in Patients with PSA Progression after Local Therapy for Prostate Cancer)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from patients who participated in E9802 and provided samples for research
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-12-07 (Actual); Primary Completion 2013-01-07 (Actual); Study Completion 2013-01-07 (Actual)

PRIMARY OUTCOMES:
PSA antibody levels are compared between baseline and follow-up at 12 weeks, as well as 24 weeks, using Wilcoxon signed-rank test | 12 weeks

SECONDARY OUTCOMES:
Concordance of PSA antibody assessment between the ECOG Immunology Laboratory and the NCI Immunology Laboratory; concordance correlation coefficient will be computed | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. DiPaola, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey